CLINICAL TRIAL: NCT02234466
Title: The Use of Preoperative Oral Dexamethasone to Improve Quality of Recovery After Breast Surgery
Brief Title: Preoperative Oral Dexamethasone to Improve Recovery After Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Faisal Siddiqui, Dr. Faisal Siddiqui, MD FRCPC, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2014:004
Record Dates: First submitted 2014-08-31; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer
Keywords: Quality of Recovery (QOR40); Breast Surgery; Clinically significant Nausea and Vomiting; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Breast Neoplasms; Vomiting; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Calcium Dobesilate; Ondansetron; Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Dexamethasone (Active Comparator): Oral dexamethasone- two 4mg tabs and one 2mg tab contained within a gelatin capsule Administered a single time, 2 hours pre-induction
  Ondansetron 6mg IV will be administered at skin closure
  Interventions: Drug: Oral dexamethasone; Drug: Ondansetron; Other: Gelatin capsule
- Gelatin pill (Placebo Comparator): Gelatin capsule contained within second gelatin capsule. Administered a single time, 2 hours pre-induction
  Ondansetron 6mg IV will be administered at skin closure
  Interventions: Drug: Ondansetron; Other: Gelatin capsule

INTERVENTIONS:
Drug: Oral dexamethasone — Patients will received their study drug ( or placebo) 2 hours pre-induction. Allowing for the shifting schedules of the OR with the possibility of the previous case finishing early or late, the allowable range is 90-200 minutes pre-induction.
  Other Names: Decadron
  Arms: Oral Dexamethasone
Drug: Ondansetron — Patients in both groups will receive 6mg IV ondansetron at time of skin closure as their standardized prophylaxis for postoperative nausea and vomiting.
  Other Names: Zofran
Other: Gelatin capsule — Gelatin capsule enclosing either dexamethasone tabs or second gelatin capsule

SUMMARY:
Randomized controlled trial of pre-operative oral dexamethasone vs placebo for the improvement of quality of recovery from surgery. The study population is limited to breast surgery patients. The investigators will also look at the effect of our intervention on post operative nausea and vomiting.

Patients will be recruited before the date of their surgery and will complete the Quality of Recovery-40 (QOR-40) questionnaire before their surgery and at 24 hours post op. They will also complete a Clinically significant nausea and vomiting score upon discharge from the post anesthesia recovery room, repeated at 24 hours post op.

DETAILED DESCRIPTION:
Design: This will be a single centre randomized, double blind, parallel-group, intention to treat, controlled trial. Patients are randomly assigned to pre-operative oral dexamethasone or placebo

Group 1: Pre-operative oral dexamethasone (10mg-2 hours pre-induction) Group 2: Placebo Sample Size: 80 patients (80% power to detect a difference of 10 points in our primary endpoint)

Study duration: 8 months

Primary endpoint: Quality of recovery at 24 hours post operation, as measured on the QoR-40 Secondary endpoints: Clinically significant nausea and vomiting on discharge from Post-Anesthesia Recovery Room (PARR) and at 24 hours.

Study hypotheses:Pre-operative oral dexamethasone will improve patient quality of recovery compared to placebo.

Secondary hypothesis: Pre-operative dexamethasone will decrease clinically significant post operative nausea and vomiting in the post anesthesia recovery room and this benefit will endure at 24 hours.

Importance: Small studies in other adult populations suggest that IV dexamethasone may improve quality of recovery. IV dexamethasone is widely used off label for postoperative nausea and vomiting (PONV) prophylaxis, oral dexamethasone has not been studied for this indication but based on the pharmacodynamics of dexamethasone, and that modulation of nucleolar transcription is likely important in dexamethasone's clinical effect; an earlier administration time is likely of benefit, this could be facilitated by an oral (vs IV) route of administration. This study will provide the preliminary support (or absence of support) for a routine, inexpensive intervention to optimize patient outcome.

Background: Single, low dose perioperative dexamethasone is safe and beneficial but common timing of administration does not maximize effectiveness. IV dexamethasone improves quality of recovery in patients undergoing laparoscopic cholecystectomy and provides a potential 1.5 mm improvement in VAS pain scores in the first 6 hours post mastectomy, which is of questionable clinical significance. A study to determine if dexamethasone improves the quality of recovery in patients undergoing breast surgery is needed in order to provide evidence for change of practices and pre-operative oral dexamethasone offers the potential for routine, low cost administration without uncomfortable side effects.

Methods: Patients will be recruited pre-operatively and contacted by telephone for preliminary consent. They will receive consent documents on the morning of surgery and be randomized at that time, they will complete a pre-operative QOR-40 and receive oral dexamethasone or placebo. During their general anaesthesia (GA) they will all receive IV Ondansetron and have their blood glucose measured 2 hours after skin incision. On discharge from PARR they will have a clinically significant nausea and vomiting scale score recorded, repeated at 24 hours post op. They will also complete the QOR-40 at 24 hours post op.

Analysis: Data will be analyzed using analysis of variance, mixed models and t-tests.

Potential Pitfalls: As the QOR-40 instrument is a survey, it is prone to inter and intra patient variability. The investigators are controlling for inter-patient variability by having patients complete the instrument before surgery to collect an individual baseline. The investigators are relying on a 25% recruitment rate of eligible patients in order to complete the study in the stated timeframe. The study has an important but narrow focus, it is not feasible to perform subgroup analysis on the small study size.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 to 80 years of age) undergoing general anesthesia for elective breast surgery (lumpectomy or mastectomy) and providing informed consent.
* American Society of Anesthesia (ASA) class I, II, & III patients

Exclusion Criteria:

* ASA class IV and V patients
* Pregnancy
* Diabetes
* History of allergy to any study medications
* Use of steroids or anti emetics within 1 month of surgery
* Chronic pain requiring opioid treatment
* History of alcohol or drug abuse (including smoking tobacco)
* Severe renal impairment (i.e. serum creatinine more than 160 umol/L)
* Poor English comprehension or psychiatric/central nervous system disturbance that would preclude completion of the QoR-40 questionnaire

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quality of recovery at Post operative day 1 (POD1) | 24 hours
  Quality of recovery as assessed by the QOR-40 will be assessed at POD1, with a baseline measure having been collected immediately pre-operatively.

SECONDARY OUTCOMES:
Post operative Nausea and Vomiting immediately post operatively | At discharge from Post Anesthesia Recovery Room, usually within 90 mins to 180 mins after surgery
  Assayed by the Clinically Significant Nausea and Vomiting Scale
Post operative Nausea and Vomiting in first 24 hours | The first 24 hours after surgery
  Post operative Nausea and Vomiting as assessed by the Clinically Significant Nausea and Vomiting scale on POD1, assessing the period from surgery until the assessment (not excluding post anesthesia recovery room)

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Siddiqui, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Science Centre, Winnipeg, Manitoba, Canada